CLINICAL TRIAL: NCT00133796
Title: A Phase II Study of the Effects of Herceptin in Patients With Locally Advanced HER-2/NEU Overexpressing Breast Cancer
Brief Title: Neoadjuvant Herceptin in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed to accrual 4/19/2006 / Study doesn't qualify for reporting.
Sponsor: Mothaffar Rimawi (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-10379
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: BREAST CANCER
Keywords: Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heceptin (Experimental): Herceptin administered to enrolled subjects
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — IV
  Other Names: Trastuzumab

SUMMARY:
The purposes of this study are to better understand how Herceptin causes tumors to become smaller and to find out how effective Herceptin, together with chemotherapy, is in treating advanced breast cancer.

DETAILED DESCRIPTION:
We want to determine the effects of Herceptin and to determine its efficacy in women with HER-2 overexpressing advanced breast cancer. The end-points will include the comparison of an array of histologic and molecular markers from sequential core biopsies of primary breast cancers of patients receiving Herceptin.

The other aim of this study would be to determine clinical response to therapy with Herceptin and Taxotere.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be female.
* Informed consent must be signed.
* Women with locally advanced breast cancers or primary breast cancers with concomitant gross metastatic disease are eligible. Locally advanced cancers must be of clinical and/or radiologic size > 4 cm, and/or are deemed surgically inoperable.
* Her2/neu overexpressing tumors defined as HercepTest score of 3+, or >/= one-third of invasive tumor showing membranous staining, or fluorescence in situ hybridization (FISH) positive.
* Negative serum pregnancy test (bHCG) within 7 days of starting study, if of child-bearing potential.
* Kidney and liver function tests - all within 1.5 times of the institution's upper limit of normal.
* Performance status (World Health Organization [WHO] scale) < 2 and life expectancy > 6 months.
* Age > 18.
* No metastatic disease without concomitant primary breast cancer.
* No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

* Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
* Severe underlying chronic illness or disease.
* Cardiomyopathy or baseline left ventricular ejection fraction (LVEF) < 50%.
* Patients on other investigational drugs while on study.
* Severe or uncontrolled hypertension defined as blood pressure (BP) > 180/100 on three separate occasions.
* History of congestive heart failure.
* History of coronary arterial disease.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-10; Primary Completion 2005-09 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The effects of Herceptin and its efficacy in women with HER-2 overexpressing advanced breast cancer | 1 year
  A comparison of histologic and molecular markers from sequential core biopsies of primary breast cancers of patients receiving Herceptin

SECONDARY OUTCOMES:
To determine clinical response to therapy with Herceptin and Taxotere | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center, Baylor College of Medicine
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No